CLINICAL TRIAL: NCT05881837
Title: A Multicenter, Randomized, Double-blind, Placebo- Parallel Controlled, Phase II Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Obese Subjects Without Diabetes
Brief Title: Efficacy and Safety of HRS9531 Injection in Obese Subjects Without Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS9531-201
Record Dates: First submitted 2023-05-17; First posted 2023-05-31 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, double-blind, placebo- parallel controlled Phase II clinical study
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Treatment group A (Experimental): HRS9531 injection
  Interventions: Drug: HRS9531 injection
- Treatment group B (Experimental): HRS9531 injection
  Interventions: Drug: HRS9531 injection
- Treatment group C (Experimental): HRS9531 injection
  Interventions: Drug: HRS9531 injection
- Treatment group D (Experimental): HRS9531 injection
  Interventions: Drug: HRS9531 injection
- Treatment group E (Placebo Comparator): HRS9531 injection Placebo
  Interventions: Drug: HRS9531 injection Placebo
- Treatment group F (Placebo Comparator): HRS9531 injection Placebo
  Interventions: Drug: HRS9531 injection Placebo
- Treatment group G (Placebo Comparator): HRS9531 injection Placebo
  Interventions: Drug: HRS9531 injection Placebo
- Treatment group H (Placebo Comparator): HRS9531 injection Placebo
  Interventions: Drug: HRS9531 injection Placebo

INTERVENTIONS:
Drug: HRS9531 injection — HRS9531 injection: dose level 1 for 32 weeks、level 2 for 20 weeks
  Arms: Treatment group A
Drug: HRS9531 injection — HRS9531 injection: dose level 2
  Arms: Treatment group B
Drug: HRS9531 injection — HRS9531 injection: dose level 3
  Arms: Treatment group C
Drug: HRS9531 injection — HRS9531 injection: dose level 4
  Arms: Treatment group D
Drug: HRS9531 injection Placebo — Placebo arm matching active arm HRS9531 injection dose level 1 for 32 weeks、HRS9531 injection level 2 for 20 weeks
  Arms: Treatment group E
Drug: HRS9531 injection Placebo — Placebo arm matching active arm HRS9531 injection dose level 2 for 32 weeks、HRS9531 injection level 2 for 20 weeks
  Arms: Treatment group F
Drug: HRS9531 injection Placebo — Placebo arm matching active arm HRS9531 injection dose level 3 for 32 weeks、HRS9531 injection level 2 for 20 weeks
  Arms: Treatment group G
Drug: HRS9531 injection Placebo — Placebo arm matching active arm HRS9531 injection dose level 4 for 32 weeks、HRS9531 injection level 2 for 20 weeks
  Arms: Treatment group H

SUMMARY:
To evaluate the efficacy and dose-response relationship of HRS9531 injection compared with placebo in reducing body weight in obese subjects without diabetes after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. Male or female subjects, 18-65 years of age at the time of signing informed consent;
3. At screening visit, 28.0 ≤BMI≤ 40.0 kg/m2;
4. Diet and exercise control for at least 3 months before screening visit, and less than 5 kg self-reported change within the last 3 months.

Exclusion Criteria:

1. Presence of - clinically significant lab or ECG results that may affect the evaluation of the efficacy or safety of the study drug at screening visit;
2. Uncontrollable hypertension;
3. PHQ-9 score ≥15;
4. Medical history or illness that affects your weight;
5. History of diabetes;
6. Acute infection, acute trauma, or medium to large surgery within 1 month prior to screening;
7. History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening;
8. Any organ-system malignancies developed within 5 years except for cured local basal cell cancer of the skin and in-situ cancer of the cervix;
9. Confirmed or suspected depression, bipolar disorder, suicidal tendencies, schizophrenia, or other serious mental illness;
10. History of alcohol and/or substance abuse or drug abuse within 1 year prior to screening;
11. Use of any medication or treatment that may have caused significant weight change within 3 months;
12. History of bariatric surgery;
13. Known or suspected hypersensitivity to trial product(s) or related products;
14. Participation in other clinical trials for any weight-loss indication within 3 months prior to screening, or participation in other clinical trials for any drug or medical device within 1 month prior to screening;
15. history of blood donation or blood loss in the 3 months before screening, or blood transfusion in the 2 months before screening;
16. Surgery is planned during the trial;
17. Mentally incapacitated or speech-impaired;
18. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method;
19. Researchers and relevant staff of the research Centre or other people directly involved in the implementation of the programme, and their immediate family members.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-10-13 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight | Week 0, Week 24
  Percentage Change from baseline in body weight after 24 weeks of treatment

SECONDARY OUTCOMES:
Proportion of subjects with weight loss of ≥5% from baseline in body weight after 24 weeks of treatment | Week 24
Proportion of subjects with weight loss of ≥10% from baseline in body weight after 24 weeks of treatment | Week 24
Change from baseline in body weight after 24 weeks of treatment | Week 0, Week 24
Change from baseline in waist circumference after 24 weeks of treatment | Week 0, Week 24
Change from baseline in BMI after 24 weeks of treatment | Week 0, Week 24
Change from baseline in blood pressure after 24 weeks of treatment | Week 0, Week 24
Change from baseline in total cholesterol after 24 weeks of treatment | Week 0, Week 24
Change from baseline in fasting plasma glucose (FPG) after 24 weeks of treatment | Week 0, Week 24
Change from baseline in glycosylated haemoglobin (HbA1c) after 24 weeks of treatment | Week 0, Week 24
Number of AEs During the Trial | Week 0 to Week 56
Percentage change in body weight | Week 0, Week 32
Proportion of Subjects with weight loss of ≥5% from baseline in body weight after 32 weeks of treatment | Week 32
Proportion of Subjects with weight loss of ≥10% from baseline in body weight after 32 weeks of treatment | Week 32
Change from baseline in body weight after 32 weeks of treatment | Week 0, Week 32
Change from baseline in waist circumference after 32 weeks of treatment | Week 0, Week 32
Change from baseline in BMI after 32 weeks of treatment | Week 0, Week 32
Change from baseline in blood pressure after 32 weeks of treatment | Week 0, Week 32
Change from baseline in total cholesterol after 32 weeks of treatment | Week 0, Week 32
Change from baseline in fasting plasma glucose (FPG) after 32 weeks of treatment | Week 0, Week 32
Change from baseline in glycosylated haemoglobin (HbA1c) after 32 weeks of treatment | Week 0, Week 32

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - The second affiliated hospital of Anhui medical university, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The people's hospital of Longhua.Shenzhen, Shenzhen, Guangdong
  - Department of Endocrinology，Sencond Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital, and College of Clinical Medicine of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Central Hospital Of Huangshi, Huangshi, Hubei
  - The Third People's Hospital of Hubei Province, Wuhan, Hubei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Lianyungang Hospital of TCM, Lianyungang, Jiangsu
  - The First People's Hospital Of Lianyungang, Lianyungang, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - North Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Second hospttoal of Shanxi medical University, Taiyuan, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xi'an Medical College, Xi'an, Xian
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided